CLINICAL TRIAL: NCT01586455
Title: A Single-Arm Study to Assess the Safety of Transplantation With Human Placental-Derived Stem-Cells Combined With Unrelated and Related Cord Blood in Subjects With Certain Malignant Hematologic Diseases and Non-Malignant Disorders
Brief Title: Human Placental-Derived Stem Cell Transplantation
Acronym: HPDSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 550; NYMC IRB L-10,733 (Other: New York Medical College)
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Adrenoleukodystrophy; Niemann-Pick Disease; Metachromatic Leukodystrophy; Wolman Disease; Krabbe's Disease; Gaucher's Disease; Fucosidosis; Batten Disease; Severe Aplastic Anemia; Diamond-Blackfan Anemia; Amegakaryocytic Thrombocytopenia; Myelodysplastic Syndrome; Acute Myelogenous Leukemia; Acute Lymphocytic Leukemia
Keywords: umbilical cord blood; stem cell transplantation; placental stem cell; inborn errors of metabolism; marrow failure; Severe Combined Immunodeficiency Disease; AML; ALL; MDS
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Adrenoleukodystrophy; Niemann-Pick Diseases; Leukodystrophy, Metachromatic; Wolman Disease; Leukodystrophy, Globoid Cell; Gaucher Disease; Fucosidosis; Neuronal Ceroid-Lipofuscinoses; Anemia, Aplastic; Anemia, Diamond-Blackfan; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Metabolism, Inborn Errors; X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): related cord blood with ≥3/6 HLA match to the patient and related HPDSC
  Interventions: Drug: Human Placental Derived Stem Cell
- Group B (Experimental): unrelated cord blood with ≥ 4/6 HLA match to the patient and unrelated HPDSC
  Interventions: Drug: Human Placental Derived Stem Cell
- Group C (Experimental): unrelated cord blood with ≥4/6 HLA match to the patient but related to HPDSC
  Interventions: Drug: Human Placental Derived Stem Cell
- Group D (Experimental): double unrelated cord blood units with ≥4/6 HLA match to patient and each other and unrelated HPDSC
  Interventions: Drug: Human Placental Derived Stem Cell

INTERVENTIONS:
Drug: Human Placental Derived Stem Cell — Infusions of thawed HPDSC to be given following UCB infusion.
  Other Names: HPDSC

SUMMARY:
The purpose of this clinical trial is to investigate the safety of human placental-derived stem cells (HPDSC) given in conjunction with umbilical cord blood (UCB) stem cells in patients with various malignant or nonmalignant disorders who require a stem cell transplant. Patients will get either full dose (high-intensity) or lower dose (low intensity) chemo- and immunotherapy followed by a stem cell transplantation with UCB and HPDSC.

ELIGIBILITY:
Inclusion Criteria:

* < 55 years of age
* Life expectancy greater than 3 months
* Lansky performance status ≥ 50% (children) or Karnofsky performance status ≥ 70% (adults) or ECOG performance status 0-2 (adults)
* DLCO > 50 percent predicted
* Left ventricular ejection fraction > 40% estimated
* Creatinine clearance or estimated GFR . 60 mL/min/1.73m2
* Serum bilirubin < 1.5x upper limit of normal
* Transaminases < 3x upper limit of normal
* Absence of uncontrolled infection
* HIV negative

Exclusion Criteria:

* Fanconi Anemia
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Uncontrolled infection
* Pregnant or breast-feeding females
* Received other investigational agents within 30 days prior to the start of the conditioning regimen

Ages: 0 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Safety | 100 days
  to evaluate the safety of human placental-derived stem cells (HPDSC) administered in conjunction with umbilical cord blood (UCB) stem cells in patients with malignant and non-malignant diseases.

SECONDARY OUTCOMES:
donor chimerism | 1 year
  donor chimerism will be assessed at set timepoints
engraftment | 1 year
Survival | 100 days and 180 days
Relapse | 100 days and 180 days
Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Denver, Colorado
  - New York Medical College, Valhalla, New York
  - University of Utah, Salt Lake City, Utah